CLINICAL TRIAL: NCT04979767
Title: Function of Circulating Exosomes in Sepsis-induced Immunosuppression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Kansas Medical Center (Other)
Collaborators: University of Kansas (Other)
Responsible Party: Principal Investigator, Nicholas Britt, Assistant Professor, University of Kansas Medical Center
Other Study IDs: STUDY#00145638
Record Dates: First submitted 2021-05-14; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Sepsis; Septic Shock; Sepsis Syndrome; Sepsis Bacterial; Sepsis, Severe; Sepsis Bacteremia
MeSH Terms: conditions — Sepsis; Shock, Septic; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole Blood, Plasma, PBMCs, Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis: I. ≥ 50 years with ≥ 2 chronic comorbidities II. Highly suspected bacterial infection based on clinical or radiologic evidence III. ≥ 2 systemic inflammatory response syndrome (SIRS) criteria IV. Actual/anticipated admission to intensive care unit (ICU) V. Anticipated length of hospital stay ≥ 5 days
- Control: I. ≥ 50 years with ≥ 2 chronic comorbidities II. No suspected bacterial infection III. Actual/anticipated admission to intensive care unit (ICU) IV. Anticipated length of hospital stay ≥ 5 days

SUMMARY:
This is a single-center prospective bio-specimen analysis and observational study aiming to define immune pathways disrupted in bacterial sepsis and to identify clinically useful biomarkers of immune status.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 50 years with ≥ 2 chronic comorbidities
* Highly suspected bacterial infection based on clinical or radiologic evidence
* ≥ 2 systemic inflammatory response syndrome (SIRS) criteria
* Actual/anticipated admission to intensive care unit (ICU)
* Anticipated length of hospital stay ≥ 5 days

Exclusion Criteria:

* Pregnancy
* Underlying immunosuppression (solid organ transplant, hematopoietic stem cell transplant, neutropenia, HIV infection, long-term corticosteroid use (≥ 20 mg prednisone equivalents for ≥ 14 days), immunosuppressants, radiation, chemotherapy, immune-modifying biologics, viral hepatitis, or systemic autoimmune diseases)
* Current immunotherapy use
* Confirmed COVID-19 infection

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized adult patients admitted to the intensive care unit with sepsis
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | From enrollment to 28 days
  All-cause mortality

SECONDARY OUTCOMES:
Hospital mortality | From enrollment until hospital discharge, up to 90 days
  All-cause mortality
90-day mortality | From enrollment to 90 days
  All-cause mortality
Length of stay | From enrollment until hospital discharge, up to 90 days
  Hospital length of stay
Duration of infection | From enrollment until resolution of SIRS, up to 90 days
  Time to resolution of infection

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas S Britt, PharmD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No